CLINICAL TRIAL: NCT00279552
Title: Can Recombinant Human Intrinsic Factor Be Used for Evaluation of the Vitamin B12 Absorption?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20030267
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2006-01-19 (Estimated); Status verified 2006-01

CONDITIONS: Vitamin B12 Deficiency
Keywords: Vitamin B12 deficiency; Vitamin B12 malabsorption; Intrinsic factor; Holotranscobalamin
MeSH Terms: conditions — Vitamin B 12 Deficiency

INTERVENTIONS:
Drug: Recombinant human intrinsic factor

SUMMARY:
Vitamin B12 is an essential nutrient for normal DNA-synthesis and must be supplied by animal products. Vitamin B12 deficiency may cause anemia and irreverible neurological damage. Laboratory tests are used for diagnosis of vitamin B12 deficiency, and following the diagnosis, the cause of the vitamin B12 deficiency has to be clarified. For years a test called Shilling's test has been used for evaluation of the vitamin B12 absorption. However, the Schilling's test is no longer easy accessible because of increasing difficulties to obtain the radioactively labeled vitamin B12 requested, and native human intrinsic factor for Schilling's test II (absorption of vitamin B12 attached to intrinsic factor) is no longer available in most countries. Recently, human intrinsic factor unsaturated with vitamin B12 has been expressed in the plant Arabidopsis thaliana. The purpose of this study was to examine whether recombinant human intrinsic factor is able to promote the uptake of vitamin B12 in patients with evident vitamin B12 deficiency.

DETAILED DESCRIPTION:
Vitamin B12 is an essential nutrient for normal DNA-synthesis and must be supplied by animal products. Vitamin B12 deficiency may cause anemia and irreverible neurological damage. Laboratory tests are used for diagnosis of vitamin B12 deficiency, and following the diagnosis, the cause of the vitamin B12 deficiency has to be clarified. For years a test called Shilling's test has been used for evaluation of the vitamin B12 absorption. However, the Schilling's test is no longer easy accessible because of increasing difficulties to obtain the radioactively labeled vitamin B12 requested, and native human intrinsic factor for Schilling's test II (absorption of vitamin B12 attached to intrinsic factor) is no longer available in most countries. Recently, human intrinsic factor unsaturated with vitamin B12 has been expressed in the plant Arabidopsis thaliana. The purpose of this study was to examine whether recombinant human intrinsic factor is able to promote the uptake of vitamin B12 in patients with evident vitamin B12 deficiency.

ELIGIBILITY:
Inclusion Criteria:

Patients suspected to have vitamin B12 deficiency defined as a plasma vitamin B12 below the reference interval (<200 pmol/L).

Exclusion Criteria:

Patients who were pregnant, nursing or not able to give written informed consent were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37
Dates: Start 2004-04; Study Completion 2004-12

PRIMARY OUTCOMES:
Change in holotrancobalamin

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, MD, Ph.D., Principal Investigator — Aarhus University Hospital
Locations (1):
- Department for Clinical Biochemistry, Aarhus, Denmark